CLINICAL TRIAL: NCT02321137
Title: A Randomized Prospective Multicenter Trial for Stroke Prevention by Surgical Occlusion of the Left Atrial Appendage in Patients Undergoing Aortic Bioprosthetic Surgery
Brief Title: Left Atrial Appendage CLOSURE for the Prevention of Thromboembolisms in Patients Undergoing Aortic Bioprosthesis Surgery
Acronym: LAA-CLOSURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); St. Antonius Hospital (Other); Landspitali University Hospital (Other)
Responsible Party: Principal Investigator, Tuomas Kiviniemi, MD, PhD, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTurku
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioAVR with surgical closure of LAA (Active Comparator): Aortic valve replacement with bioprosthesis according to indications in the current guidelines for the management of valvular heart disease including surgical closure of left atrial appendage
  Interventions: Procedure: Surgical closure of left atrial appendage
- BioAVR alone (Placebo Comparator): Aortic valve replacement with bioprosthesis according to indications in the current guidelines for the management of valvular heart disease.
  Interventions: Procedure: No closure of left atrial appendage

INTERVENTIONS:
Procedure: Surgical closure of left atrial appendage — aortic valve replacement with bioprosthesis according to indications in the current guidelines for the management of valvular heart disease. The operation as well as the pre and post-operative care will be performed according to local surgical policies.
  Arms: BioAVR with surgical closure of LAA
Procedure: No closure of left atrial appendage — aortic valve replacement with bioprosthesis according to indications in the current guidelines for the management of valvular heart disease.
  Arms: BioAVR alone

SUMMARY:
The primary purpose of the LAA-CLOSURE trial is to assess the efficacy and safety of surgical closure of LAA in patients undergoing aortic valve replacement. This randomized, prospective, open-label international multicenter trial will enroll 1040 patients undergoing aortic valve replacement with CHA2DS2-VASC score ≥2 but without an indication for anticoagulation at the time of enrollment. Patients will be randomized in 1:1 fashion to standard therapy + surgical closure of LAA vs. standard therapy alone. The duration of the study is five years (plus additional 10 years).

DETAILED DESCRIPTION:
Previous studies have concluded that ≥90% of AF related left atrial thrombi are located in the left atrial appendage (LAA). Surgical closure of LAA can be performed using ligation, stapler or other devices designed for this purpose during cardiac surgery. However, current evidence for surgical closure of LAA is scarce and no large scale randomized prospective clinical trials addressing this issue have been published. American College of Cardiology (ACC)/ American Heart Association (AHA) guidelines state that LAA exclusion should be considered in patients with recurrent and persistent AF who remain symptomatic with heart rate control and where antiarrhythmic medication is not tolerated or no longer effective. Current European Association of Cardiothoracic Surgery (EACTS) guidelines conclude that there is no proven benefit of surgical LAA exclusion in terms of stroke reduction or mortality benefit (level of evidence 2a B), and if exclusion is contemplated, devices designed for appendage exclusion should be used rather than a cut-and-sew or stapling technique. These guidelines are based on small poorly designed descriptive trials and only one small randomized trial.

LAA-CLOSURE trial aims to assess efficacy and safety of prophylactic surgical closure of LAA in patients undergoing aortic valve replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing aortic valve replacement (+/- coronary bypass AND/OR mitral valve surgery) according to clinical indications (ESC guidelines for the management of valvular heart disease)
2. Age ≥18 years
3. No indication for long term anticoagulation at the time of enrollment.
4. Patients with CHADS-VASC score ≥2
5. Patient is willing to comply with specified follow-up evaluations
6. Patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written informed consent, approved by the appropriate Medical Ethics committee or Institutional Review Board.

Exclusion Criteria:

* Age < 18 years
* Expected survival < 1 year
* Chronic atrial fibrillation
* Indication for long term anticoagulation therapy before the index procedure
* Mechanical valve implantation previously or at the index procedure
* Any significant medical condition, which in the Investigator's opinion may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-04-30 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
A composite of stroke, systemic embolism and cardiovascular mortality | 5 years

SECONDARY OUTCOMES:
stroke/systemic embolism | 5 years
cardiovascular mortality | 5 years
Net adverse events (primary endpoint and major bleeding) | 5 years
Hospitalization for decompensated heart failure | 5 years
Major bleeding (BARC 3a, b, c or 5) | 5 years
Any bleeding (BARC 1, 2 3a, b, c or 5) | 5 years
Surgery related bleeding (BARC 4) | 5 years
Stroke | 30 days postoperatively
  30D Post-op thromboembolism
A composite outcome of any of the following: stroke, systemic embolism and cardiovascular mortality | 30 days postoperatively
  A composite outcome of stroke, systemic embolism and cardiovascular mortality

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Kiviniemi, MD, PhD, Principal Investigator — Turku University Hospital, Turku, Finland
Locations (4):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku
- St Antonius Hospital, Utrecht, Netherlands

REFERENCES:
- See also: Published trial protocol — https://doi.org/10.1016/j.ahj.2021.03.014